CLINICAL TRIAL: NCT06626113
Title: Concomitantly Higher Resting Arterial Blood Pressure and Transduction of Sympathetic Neural Activity in Human Obesity Without Hypertension
Brief Title: Transduction of Sympathetic Neural Activity in Human Obesity Without Hypertension
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: VITAMINC
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Ascorbic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Obese
  Interventions: Drug: ascorbic acid

INTERVENTIONS:
Drug: ascorbic acid — ascorbic acid

SUMMARY:
In addition to chronically elevated MSNA, there is a growing recognition that hypertension in states of insulin resistance and obesity may also be attributed to an increased vascular sensitivity to MSNA (1, 2, 13, 36-38). To study this phenomenon, we quantify vascular sensitivity to MSNA using an innovative, moment-to-moment assessment of the blood pressure response following individual bursts of muscle sympathetic nerve activity (MSNA), (10, 11, 34, 37). This approach is termed 'sympathetic-vascular transduction (SVT).' We will examine the hypothesis that SVT is exaggerated in obesity and insulin resistance and is attenuated by suppression of oxidative stress. Oxidative stress is the overabundance of reactive oxygen species and is another hallmark of hypertension, obesity, and insulin resistance. Oxidative stress can be safely reduced via intravenous infusion of ascorbic acid (Vit C) (4, 28). Therefore, we will use a randomized, double-blinded, placebo-controlled approach to test the hypothesis that elevated SVT will be attenuated by suppression of oxidative stress via ascorbic acid I.V. infusion compared with saline I.V. infusion (placebo) in obese adults with insulin resistance. Our study will identify a unique mechanism that can be targeted to reduce the excessively high prevalence of hypertension and risk for CVD in obesity and insulin resistance.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo-controlled study. Eligible participants will have a total of 3 visits to the laboratory. At the first experimental visit individuals will be randomized in a double-blind fashion to either ascorbic acid or placebo and the alternative treatment will be given on the subsequent study visit. The KU Investigational Pharmacy will perform the blinded randomization.

1. Week 1 Visit 1 Screening
2. Week 2 Visit 2 Randomization and Experimental visit
3. Week 5 Visit 3 Experimental visit

ELIGIBILITY:
Inclusion criteria:

1. Obese: BMI >25 m/kg2
2. Elevated insulin resistance: HOMA-IR > 2.5 (calculation based on fasting glucose and insulin concentrations in blood)
3. Middle-aged: 35-65 years
4. Participants must be willing and able to discontinue taking any vitamin C or E supplements or omega-3 fatty acids beginning 2 weeks prior.
5. Able and willing to provide written informed consent

Exclusion criteria:

1. Currently taking a statin or antihypertension medication
2. Hyperlipidemia: Fasting triglycerides < 250 mg/dL
3. Hypertension: >130/80 mmHg
4. History of heart disease (e.g., myocardial infarction, stent)
5. History of vascular disease (e.g., bypass, stroke)
6. Individuals with narrow angle glaucoma

   -

Ages: 18 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — self-reported
Study Population: Obese
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Sympathetic transduction | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States